CLINICAL TRIAL: NCT04737486
Title: A Randomized, Double-blind, Placebo-controlled Phase 1 Single and Multiple-Dose Pharmacokinetic First-in-Human Study of AV-001 in Healthy Subjects
Brief Title: A First-in-Human Study of AV-001 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vasomune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV001-PK-001
Record Dates: First submitted 2020-12-31; First posted 2021-02-03 (Estimated); Last update posted 2021-03-24 (Actual); Status verified 2021-01

CONDITIONS: Covid19-associated ARDS; Covid19; ARDS
Keywords: Vascular normalization; Endothelial stability
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Single and multiple ascending dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Single Ascending Dose Cohort 1-4 (Experimental): Intervention: AV-001, 6 subjects per cohort will receive single doses of 1.4 µg/kg up to 56 µg/kg of AV-001 by intravenous bolus injection.
  Interventions: Drug: AV-001
- Single Ascending Dose Cohort 1-4, Placebo (Placebo Comparator): Intervention: Placebo, 2 subjects per cohort will receive single doses of D-PBS placebo by intravenous bolus injection.
  Interventions: Other: Placebo
- Multiple Ascending Dose Cohort 1-2 (Experimental): Intervention: AV-001, 6 subjects per cohort will receive multiple doses of 1.4 µg/kg/day up to 56 µg/kg/day of AV-001 daily for 7 consecutive days by intravenous bolus injection.
  Interventions: Drug: AV-001
- Multiple Ascending Dose Cohort 1-2, Placebo (Placebo Comparator): Intervention: Placebo, 2 subjects per cohort will receive multiple doses of D-PBS placebo daily for 7 consecutive days by intravenous bolus injection.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AV-001 — AV-001 (mpaBr) Cl for Injection 2.5 mg/mL
  Arms: Multiple Ascending Dose Cohort 1-2; Single Ascending Dose Cohort 1-4
Other: Placebo — D-PBS
  Arms: Multiple Ascending Dose Cohort 1-2, Placebo; Single Ascending Dose Cohort 1-4, Placebo

SUMMARY:
Phase 1 randomized, double-blind, placebo-controlled single ascending dose (SAD) and multiple ascending dose (MAD) first-in-human study in healthy subjects. Safety and tolerability assessments will be conducted, and blood samples will be taken pre-dose and at several time points post-dose for pharmacokinetic (PK) and pharmacodynamics (PD) analysis.

DETAILED DESCRIPTION:
In the SAD segment of the study, up to 4 ascending cohorts of 8 healthy subjects each will receive a single dose of study drug (AV-001 or placebo) in a sequential ascending manner. Planned doses may be adapted depending on emergent safety, tolerability and available PK data. Screening evaluations will occur from Day -28 to Day -2. Eligible subjects will be admitted to the clinical unit on Day -2. On Day 1, subjects will be randomized to AV-001 (6 subjects) or placebo (2 subjects) and receive a single dose of study drug. Subjects will be discharged on Day 2 after all post dose assessments have been completed and if there are no medical reasons for a longer stay in the clinical unit. An end of study visit will be conducted 7 to 10 days after Day 1 or at early termination.

An initial sentinel group consisting of 1 subject receiving AV-001 and 1 subject receiving placebo will proceed for each cohort prior to treatment of the remainder of the cohort. After study drug administration to the sentinel group and an appropriate safety interval (at least 24 hours and per the discretion of the Principal Investigator (PI)), the remaining 5 subjects will receive a single dose of AV-001 and 1 subject will receive placebo administered in the same manner.

PK blood samples will be collected at 15 time points relative to study drug dosing on Day 1. PD blood samples for will be collected at 6 time points on Day 1.

In the MAD segment of the study, up to 2 ascending cohorts of 8 subjects each will receive once daily doses of study drug (AV-001 or placebo) for at least 7 days in a sequential ascending manner. Planned doses may be adapted and will be determined by the safety, tolerability and PK data from the SAD part of the study. Screening evaluations will occur from Day -28 to Day -2. Eligible subjects will be admitted to the clinical unit on Day -2. On Day 1, subjects will be randomized to AV-001 (6 subjects) or placebo (2 subjects). Subjects will receive once-daily doses of study drug from Day 1 through Day 7. Subjects will be discharged on Day 8 after all post dose assessments have been completed and if there are no medical reasons for a longer stay in the clinical unit. An end of study visit will be conducted 7 to 10 days after Day 7 or at early termination.

PK blood samples will be collected at 15 time points relative to study drug dosing on Day 1 and Day 7 in addition to predose levels on Days 2 to 6. PD blood samples for will be collected at 6 time points on Day 1 and Day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Subject voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB) approved informed consent prior to performing any of the Screening Visit procedures
2. Males and female subjects of nonchildbearing potential between 18 to 65 years of age, inclusive, at the Screening Visit
3. Male subjects must agree to use a highly effective form of contraception (e.g., abstinence, double-barrier methods, have had a vasectomy or have sexual partner(s) of nonchildbearing potential) at the time of the Screening Visit and for 30 days after the dose or last dose of IMP. Male subjects must also agree to not donate sperm for the duration of the study and until 90 days after the dose or last dose of IMP
4. Female subjects must be nonpregnant and nonlactating and either surgically sterile (e.g., bilateral tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or postmenopausal for > 12 months. Postmenopausal status will be confirmed through testing of follicle-stimulating hormone (FSH) levels ≥ 40 U/mL at the Screening Visit for amenorrheic female subjects
5. Non smokers (or other nicotine use) as determined by history (no nicotine use over the past three months) and by negative urine cotinine concentration at the Screening Visit and admission
6. Body weight > 50 kg and <150 kg at the Screening Visit
7. Body mass index (BMI) between 19 and 32 kg/m2, inclusive, at the Screening Visit
8. Vital sign measurements at the Screening Visit and on Day 1 within the following ranges (measurements may be repeated once per the discretion of the Principal Investigator):

   1. Systolic blood pressure: 110 to 139 mmHg
   2. Diastolic blood pressure: 70 to 89 mmHg
   3. Pulse rate: 40 to 90 bpm
   4. Oral body temperature: 35.0°C to 37.5°C A subject should not be included if their standing vital signs (relative to sitting) show findings which, in the opinion of the Principal Investigator, are associated with the clinical manifestation of postural hypotension (i.e., absence of any other cause). These changes include either a > 20 mmHg decrease in systolic, a >10 mmHg decrease in DBP, a > 30 bpm increase in heart rate from sitting to standing or > 120 bpm
9. Healthy, determined by prestudy medical evaluation (medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory evaluations)

Exclusion Criteria:

1. Subject has clinically significant history or evidence of cardiovascular, hematologic, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological or psychiatric disorder(s) as determined by the Principal Investigator or designee
2. Subject has any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs, in the opinion of the Principal Investigator
3. Subject has a history of autonomic dysfunction (e.g., a history of fainting, orthostatic hypotension)
4. Subject has any concurrent disease or condition that, in the opinion of the Principal Investigator, would make the subject unsuitable for participation in the clinical study
5. Subject has history of alcohol and/or illicit drug abuse within 2 years of entry
6. Subject has positive test for hepatitis B surface antigen (HBsAg), hepatitis C antibody (anti-HCV) or human immunodeficiency virus (HIV) type 1 and 2 antibodies
7. Subject has positive breath alcohol test for ethanol at the Screening Visit or admission.
8. Subject has positive urine drug test at the Screening Visit or admission
9. Female subjects are breastfeeding or female subjects with a positive serum pregnancy test at the Screening Visit or admission
10. Subject is unwilling to avoid consumption of xanthine containing products (e.g., caffeine in coffee, tea, chocolate) within 48 hours prior to admission until discharge from the clinical site
11. Subject is unwilling to avoid use of alcohol or alcohol-containing foods, medications or beverages, within 48 hours prior to admission until discharge from the clinical site
12. Subject has donated blood (> 500 mL) or blood products within 2 months (56 days) prior to admission
13. Subject has used over-the-counter (OTC) medications (including vitamins), 7 days prior to admission or prescription medications or herbal remedies from 14 days prior to admission until the End-of-Study Visit. By exception, paracetamol/acetaminophen ≤ 1000 mg per day and hormonal replacement therapy are permitted
14. Subject has participated in a clinical study or used an investigational drug within 30 days or 5 × half lives (whichever is the longer interval) prior to the Screening Visit
15. Subject is unwilling to abstain from vigorous exercise from 48 hours prior to admission until the End of Study Visit
16. Subject has a history of hypersensitivity to the study drug or any of the excipients or to medicinal products with similar chemical structures or containing PEG (i.e., GripaNait® cough syrup, Betadine® antiseptic solution/cream)
17. Subject is unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope and possible consequences of the clinical study
18. Subject is unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up visits and improbability of completing the clinical study
19. Subject has a positive test result for SARS-CoV-2 before randomization
20. Subject has previously been enrolled in this clinical study
21. Vulnerable subjects defined as individuals whose willingness to volunteer in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate (e.g., persons in detention, minors and those incapable of giving consent)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Participants experiencing drug-related adverse events | 8 days following a single intravenous dose (SAD) or 8 days following 7 consecutive daily intravenous doses (MAD)
  Number of drug-related adverse events as determined by abnormal clinical laboratory tests, vitals signs, continuous blood pressure monitoring and collection (systolic, diastolic, pulse pressure, heart rate and mean arterial pressure), physical exam and ECG parameters

SECONDARY OUTCOMES:
Cmax: Maximum plasma AV-001 concentration | 1 day following a single intravenous dose (SAD); 8 days following 7 consecutive daily intravenous doses (MAD)
  Maximum plasma AV-001 concentration
Tmax: Time of maximum plasma AV-001 concentration | 1 day following a single intravenous dose (SAD); 8 days ollowing 7 consecutive daily intravenous doses (MAD)
  Time of maximum plasma AV-001 concentration
AUClast: AUC from predose (time 0) to the time of the last quantifiable concentration | 1 day following a single intravenous dose (SAD); 8 days following 7 consecutive daily intravenous doses (MAD)
  AUC from predose (time 0) to the time of the last quantifiable concentration
AUCinf: AUC from predose (time 0) extrapolated to infinite time | 1 day following a single intravenous dose (SAD); 1 day following first daily intravenous dose (MAD)
  AUC from predose (time 0) extrapolated to infinite time
AUCtau: AUC over the dose interval time | 8 days following 7 consecutive daily intravenous doses (MAD)
  AUC over the dose interval time
λz: The terminal elimination rate | 1 day following a single intravenous dose (SAD); 8 days following 7 consecutive daily intravenous doses (MAD)
  The terminal elimination rate
T½: Terminal elimination half-life | 1 day following a single intravenous dose (SAD); 8 days following 7 consecutive daily intravenous doses (MAD)
  Terminal elimination half-life
CL: Total body clearance | 1 day following single intravenous dose (SAD); 8 days following 7 consecutive daily intravenous doses (MAD)
  Total body clearance
Vz: Apparent volume of distribution | 1 day following a single intravenous dose (SAD); 8 days following 7 consecutive daily intravenous doses (MAD)
  Apparent volume of distribution
Ctau: Trough plasma concentration | 6 days (day 2 through day 6 of daily intravenous doses) (MAD)
  Trough plasma concentration
Rac(AUCtau), Rac(Cmax), Rac(Ctau): Accumulation ratios assessment | 8 days following 7 consecutive daily intravenous doses (MAD)
  Accumulation ratios assessment
LM: Time-invariance ratio calculation | 8 days following 7 consecutive daily intravenous doses (MAD)
  Time-invariance ratio calculation

CONTACTS AND LOCATIONS:
Overall Officials: Leela Vrishabhendra, MD, Principal Investigator — Medpace, Inc.
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States